CLINICAL TRIAL: NCT03262753
Title: LOVE-COARCT Study: Long-term Outcomes and Vascular Evaluation After Coarctation of the Aorta Treatment
Brief Title: Long-term Outcomes and Vascular Evaluation After Coarctation of the Aorta Treatment
Acronym: LOVE-COARCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Collaborators: Centro de Estudos de Doenças Crónicas (Other); Baylor College of Medicine (Other); Lucile Packard Children's Hospital (Other); Children's Hospital Colorado (Other); University of Nebraska (Other); Boston Children's Hospital (Other); Instituto Superior Técnico de Lisboa (Unknown); Caselas, Ressonância Magnética, S.A. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHLC.CI.69.2012
Record Dates: First submitted 2017-08-08; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Aortic Coarctation; Arterial Stiffness; PULSE WAVE VELOCITY; Functional Magnetic Resonance Imaging; Vascular Endothelium
MeSH Terms: conditions — Aortic Coarctation | interventions — Surgical Procedures, Operative; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- surgery: Primary end-to-end surgical treatment of coarctation of the aorta
  Interventions: Procedure: Surgery
- balloon dilation: Primary balloon dilation treatment of coarctation of the aorta
  Interventions: Procedure: Balloon dilation
- stent: Primary stent dilation treatment of coarctation of the aorta
  Interventions: Procedure: Stent

INTERVENTIONS:
Procedure: Surgery — Primary end-to-end surgical treatment of coarctation of the aorta
  Groups: surgery
Procedure: Balloon dilation — Primary balloon dilation treatment of coarctation of the aorta
  Groups: balloon dilation
Procedure: Stent — Primary stent dilation treatment of coarctation of the aorta
  Groups: stent

SUMMARY:
Background: Coarctation of the aorta (CoA) can be treated using surgery, balloon angioplasty or stent implantation. Although short-term results are excellent with all three treatment modalities, long term cardiovascular (CV) morbidity and mortality remain high, likely due to persistently abnormal vascular function. The effects of treatment modality on long term vascular function remain uncharacterized. The goal of this study is to assess vascular function in this patient population for comparison among the treatment modalities. Methods: Vascular function in large and small arteries will be prospectively assessed fusing multiple non-invasive modalities, and the results will be compared among the three groups of CoA patients previously treated using surgery, balloon angioplasty or stent implantation after frequency matching for confounding variables. A comprehensive vascular function assessment protocol was created to be used in 7 centers. The primary outcome is arterial stiffness measured by arterial tonometry. Inclusion and exclusion criteria were carefully established after consideration of several potential confounders. Sample size was calculated for the primary outcome variable. Conclusions: Treatment modalities for CoA may have distinct impact on large and small arterial vascular function. The results of this study will help identify the treatment modality that is associated with the most optimal level of vascular function, which, in the long term may reduce CV risk.

DETAILED DESCRIPTION:
Study overview. This cross-sectional prospective observational study of patients with CoA previously treated using one of three treatment modalities assesses if treatment type is associated with differences in vascular function. The three treatment groups will be frequency-matched for key confounding variables.

Study feasibility. The investigators assembled a multi-disciplinary team with proven expertise in epidemiology, clinical trial design, congenital heart disease, non-invasive imaging, interventional cardiology, vascular function assessment, preventive cardiology and statistical analysis. A multicenter design is used to ensure sufficient statistical power in evaluating the hypothesis.

Participating centers and study core laboratories. Patients are recruited at six large pediatric cardiac centers from Portugal and USA.

Screening procedures. The medical records of potentially eligible patients are screened by a local study investigator using a pre-specified screening form to ensure that they satisfy our selection criteria.

Overview of the study workflow. Study procedures will occur in a one- or two-day visit. Upon arrival for testing, formal consent for participation will be obtained. Assessment of arterial stiffness, endothelial function, and blood sampling for biomarkers will be done while fasting. Cardiopulmonary stress test will be performed on the same day. CMR and ambulatory blood pressure monitoring (ABMP) will be arranged for the same or for the following day. When the study tests cannot be completed at the first visit, they will be completed within 3 months of the first visit. The study protocol was approved by the Institutional Review Board or Institutional Ethics Committee at each participating center, and informed consent and assent will be obtained, depending on age, from patients and their parents/legal guardians before trial enrollment.

Recruitment. A review of the patient database at each participating institution will be performed to assemble a cohort of patients with CoA who have previously undergone treatment with balloon dilation, surgery or stenting. Study data will be collected and managed using REDCap electronic data capture tools hosted at Boston Children's Hospital.

Data collection. A retrospective chart review will be performed to collect demographic and clinical data including severity of coarctation, type and details of CoA treatment and presence of associated conditions.

Diagnostic procedures.

Arterial Stiffness Plan & Rationale:

Measurements: Carotid-femoral PWV (cfPWV) will be measured using applanation tonometry. Segmental PWV is measured using CMR. Segmental measures of arterial distensibility will be measured using CMR. Other parameters that describe arterial stiffness reflect the relationship of arterial change in diameter to change in pressure and include aortic strain (relative change in diameter), compliance (absolute change in diameter in response to a change in pressure), distensibility (relative change in diameter in response to a change in pressure), and the aortic stiffness β index (distensibility using the logarithmic conversion of the relative pressure). Applanation tonometry, which uses a probe or tonometer to record the pulse wave with a transducer, is the most widely accepted method for estimating PWV and both the NIHem (Cardiovascular Engineering, Inc., Norwood, MA USA) and the SphygmoCor (AtCor Medical, West Ryde, NSW, Australia) devices have been validated in large cohort trials. Both devices will be used, based on local availability.

Endothelial Function Measurements: Endothelium-dependent reactive hyperaemia index and augmentation index will be measured using the EndoPAT 2000 system (Itamar Medical, Caesarea, Israel). The protocol includes measures to minimize the influence of the autonomic nervous system.

Pulse Waveform Analysis: Central aortic pressure and pulse pressure will be measured using applanation tonometry). Augmentation index will be measured using applanation tonometry and Endo-PAT. CAP, PP and AIx can be measured non-invasively using radial or carotid applanation tonometry (and Endo-PAT for AIx), calibrated by the peripheral diastolic and mean arterial pressure. Both the NIHem system and the SphygmoCor device were used.

Blood Pressure Phenotype will be measured using conventional standard techniques including auscultatory right arm BP measurement, measurement of BP gradient between arm and leg, BP response during treadmill exercise stress testing (ET) and ABPM. Based on the auscultatory BP and ABPM results, the appropriate children and adult guidelines will be used to classify patients. Patients currently on antihypertensive medication will be classified as hypertensive.

Biomarkers: The researchers will measure biomarkers of endothelial function (total oxides of nitrogen- NOx and ADMA), inflammation (hs-CRP), vascular wall function (VCAM-1 and IL-1β) and vascular remodeling (MMP-2; MMP-9 and TGF-beta1). NOx will be determined by chemiluminescence (Sievers NOAnalyzer 280i) and all remaining measurements will be performed with appropriate enzyme-linked immunosorbent assay (ELISA) kits: ADMA (Sunred Biological Technology, Shanghai, China); hs-CRP (BoosterBio, Pleasanton, USA); VCAM-1; IL-1β; MMP-9; MMP-2 and TGFβ-1 (RayBiotech, Inc. Norcross, USA).

Left Ventricular Mass Assessment by CMR. The altered blood pressure phenotype that persists after CoA treatment represents an increase in afterload that leads to LV hypertrophy. Our CMR protocol will include sequences that allow this quantification.

Cardiovascular Health Assessment: The researchers will assess health factors (blood pressure, total cholesterol, plasma glucose), behaviors (smoking, body mass index BMI, physical activity and diet) and family history of cardiovascular disease and risk factors. A questionnaire was implemented to assess family history of CV disease and ICVH according to the procedures and recommendations of the American Heart Association.

Statistical Considerations. The treatment groups will be frequency-matched for documented confounders. The confounding variables will include: (a) Age at treatment; (b) Current age; (c) Bicuspid aortic valve as it is associated with impaired aortic elasticity. Because of the relatively large number of matching variables and three treatment groups, matching individual subjects was not feasible. During analysis, the treatment groups will be compared for each of these confounding variables and appropriate adjustments made, if needed. Differences in the confounding variables across the three treatment groups will be evaluated using Fisher's exact test for severity of coarctation and the Kruskal-Wallis test for age at treatment, current age and bicuspid aortic valve. The primary outcome variable will be carotid-femoral PWV assessed by tonometry. Differences in cfPVW across groups will be explored using one-way analysis of variance. If differences in matching variables are detected among the groups, adjustment will be made using analysis of covariance. Post-hoc analyses will be performed as necessary.

Sample size estimates were obtained based on prior data that show that ascending- descending PWV measured by CMR is 3.3±0.6 m/s in normal subjects and 4.7±1.1 m/sec after CoA surgery.22, 70 Sample size estimates for comparison of PVW between three equal sized treatment groups (assuming overall significance level=0.05 and power=0.8) are shown in table 2. The investigators plan on recruiting 24 to 30 patients in each group for a total sample size of 72 to 90.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of isthmic coarctation of the aorta;
* Current age between 8 (to allow cooperation with study procedures) and 35 years (to avoid confounding by aging-related vascular dysfunction); and
* Treatment for CoA after 1994, after which all three modalities were in clinical use.

Exclusion Criteria:

* Residual CoA defined by a systolic upper-to-lower extremity BP gradient> 20mmHg;
* Co-morbidities that may independently affect vascular function, including associated significant congenital heart disease, history of known vasculopathy, genetic syndromes or other cardiovascular risk factors;
* History of two treatment types for CoA; and
* CoA types likely representing a different entity or patients amenable to one single treatment type (surgery), including atypical CoA site (such as mid-thoracic or abdominal), severe hypoplasia of the aortic arch, and an age of treatment <1 year of age.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with isthmic coarctation of the aorta, treated after 1994, submitted to only one of either of the three procedures described above.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Vascular function | 6 months to 35 years after primary treatment
  Arterial stiffness assessed with carotid-femoral PWV measurements by tonometry

SECONDARY OUTCOMES:
Cardiac Magnetic Resonance functional indexes | 6 months to 35 years after primary treatment
  Ascending-descending aorta PWV and aorta strain, distensibility, compliance and aortic stiffness β index measured by CMR
Endothelial function | 6 months to 35 years after primary treatment
  Endothelial function determined by endothelial pulse amplitude testing
Pulse wave form | 6 months to 35 years after primary treatment
  Pulse wave form analysis using arterial tonometry
Blood pressure phenotype | 6 months to 35 years after primary treatment
  Blood pressure phenotype at rest, during ambulatory measurement, and at peak exercise
Left ventricular mass | 6 months to 35 years after primary treatment
  Left ventricular mass assessed by Cardiac Magnetic Resonance
Left ventricular systolic function | 6 months to 35 years after primary treatment
  Left ventricular systolic function assessed by Cardiac Magnetic Resonance
Biomarkers of endothelial function | 6 months to 35 years after primary treatment
  biomarkers of endothelial function (total oxides of nitrogen- NOx and ADMA),
Biomarkers of vascular inflammation | 6 months to 35 years after primary treatment
  biomarkers of inflammation (hs-CRP).
Biomarkers of vascular wall function | 6 months to 35 years after primary treatment
  biomarkers of vascular wall function (VCAM-1 and IL-1β)
Biomarkers of vascular remodeling | 6 months to 35 years after primary treatment
  biomarkers of vascular remodeling (MMP-2; MMP-9 and TGF-beta1).

CONTACTS AND LOCATIONS:
Overall Officials: José D Martins, MD MSc, Principal Investigator — Centro Hospitalar de Lisboa Central; Miguel Mota Carmo, MD PhD, Study Chair — Centro de Estudos de Doenças Crónicas da Faculdade de Ciências Médicas da Universidade Nova de Lisboa
Locations (1):
- Department of Pediatric Cardiology, Hospital de Santa Marta, Centro Hospitalar de Lisboa Central, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Trends in infant mortality attributable to birth defects--United States, 1980-1995. MMWR Morb Mortal Wkly Rep. 1998 Sep 25;47(37):773-8. PMID 9769135
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Background] Prakash A, Adlakha H, Rabideau N, Hass CJ, Morris SA, Geva T, Gauvreau K, Singh MN, Lacro RV. Segmental Aortic Stiffness in Children and Young Adults With Connective Tissue Disorders: Relationships With Age, Aortic Size, Rate of Dilation, and Surgical Root Replacement. Circulation. 2015 Aug 18;132(7):595-602. doi: 10.1161/CIRCULATIONAHA.114.014934. Epub 2015 Jun 25. PMID 26115544
- [Background] Takagi H, Manabe H, Kawai N, Goto SN, Umemoto T. Circulating matrix metalloproteinase-9 concentrations and abdominal aortic aneurysm presence: a meta-analysis. Interact Cardiovasc Thorac Surg. 2009 Sep;9(3):437-40. doi: 10.1510/icvts.2009.208835. Epub 2009 Jun 12. PMID 19525292
- [Background] Barbaro NR, Fontana V, Modolo R, De Faria AP, Sabbatini AR, Fonseca FH, Anhe GF, Moreno H. Increased arterial stiffness in resistant hypertension is associated with inflammatory biomarkers. Blood Press. 2015 Feb;24(1):7-13. doi: 10.3109/08037051.2014.940710. Epub 2014 Jul 25. PMID 25061978
- [Background] Forbes TJ, Kim DW, Du W, Turner DR, Holzer R, Amin Z, Hijazi Z, Ghasemi A, Rome JJ, Nykanen D, Zahn E, Cowley C, Hoyer M, Waight D, Gruenstein D, Javois A, Foerster S, Kreutzer J, Sullivan N, Khan A, Owada C, Hagler D, Lim S, Canter J, Zellers T; CCISC Investigators. Comparison of surgical, stent, and balloon angioplasty treatment of native coarctation of the aorta: an observational study by the CCISC (Congenital Cardiovascular Interventional Study Consortium). J Am Coll Cardiol. 2011 Dec 13;58(25):2664-74. doi: 10.1016/j.jacc.2011.08.053. PMID 22152954
- [Background] Brown ML, Burkhart HM, Connolly HM, Dearani JA, Cetta F, Li Z, Oliver WC, Warnes CA, Schaff HV. Coarctation of the aorta: lifelong surveillance is mandatory following surgical repair. J Am Coll Cardiol. 2013 Sep 10;62(11):1020-5. doi: 10.1016/j.jacc.2013.06.016. Epub 2013 Jul 10. PMID 23850909
- [Background] Martins JD, De Sousa L, Matos P, Pinto FF. Percutaneous closure of a large coronary fistula. Rev Port Cardiol. 2009 Sep;28(9):1017-8. No abstract available. PMID 19998812
- [Background] Hager A, Kanz S, Kaemmerer H, Schreiber C, Hess J. Coarctation Long-term Assessment (COALA): significance of arterial hypertension in a cohort of 404 patients up to 27 years after surgical repair of isolated coarctation of the aorta, even in the absence of restenosis and prosthetic material. J Thorac Cardiovasc Surg. 2007 Sep;134(3):738-45. doi: 10.1016/j.jtcvs.2007.04.027. PMID 17723827
- [Background] Bocelli A, Favilli S, Pollini I, Bini RM, Ballo P, Chiappa E, Zuppiroli A. Prevalence and long-term predictors of left ventricular hypertrophy, late hypertension, and hypertensive response to exercise after successful aortic coarctation repair. Pediatr Cardiol. 2013 Mar;34(3):620-9. doi: 10.1007/s00246-012-0508-0. Epub 2012 Sep 30. PMID 23052661
- [Background] Meyer AA, Joharchi MS, Kundt G, Schuff-Werner P, Steinhoff G, Kienast W. Predicting the risk of early atherosclerotic disease development in children after repair of aortic coarctation. Eur Heart J. 2005 Mar;26(6):617-22. doi: 10.1093/eurheartj/ehi037. Epub 2004 Dec 16. PMID 15618050
- [Background] Lam YY, Mullen MJ, Kaya MG, Gatzoulis MA, Li W, Henein MY. Left ventricular long axis dysfunction in adults with "corrected" aortic coarctation is related to an older age at intervention and increased aortic stiffness. Heart. 2009 May;95(9):733-9. doi: 10.1136/hrt.2008.158287. Epub 2008 Dec 18. PMID 19095712
- [Background] Shang Q, Sarikouch S, Patel S, Schuster A, Steinmetz M, Ou P, Danford DA, Beerbaum P, Kutty S. Assessment of ventriculo-vascular properties in repaired coarctation using cardiac magnetic resonance-derived aortic, left atrial and left ventricular strain. Eur Radiol. 2017 Jan;27(1):167-177. doi: 10.1007/s00330-016-4373-8. Epub 2016 May 23. PMID 27215582
- [Background] Mizia-Stec K, Trojnarska O, Szczepaniak-Chichel L, Gabriel M, Bartczak A, Cieplucha A, Chudek J, Grajek S, Tykarski A, Gasior Z. Asymmetric dimethylarginine and vascular indices of atherosclerosis in patients after coarctation of aorta repair. Int J Cardiol. 2012 Jul 26;158(3):364-9. doi: 10.1016/j.ijcard.2011.01.037. Epub 2011 Feb 18. PMID 21334083
- [Background] Brili S, Tousoulis D, Antoniades C, Aggeli C, Roubelakis A, Papathanasiu S, Stefanadis C. Evidence of vascular dysfunction in young patients with successfully repaired coarctation of aorta. Atherosclerosis. 2005 Sep;182(1):97-103. doi: 10.1016/j.atherosclerosis.2005.01.030. Epub 2005 Feb 24. PMID 16115479
- [Background] Jesus CA, Assef JE, Pedra SR, Ferreira WP, Davoglio TA, Petisco AC, Saleh MH, Le Bihan DC, Barretto RB, Pedra CA. Serial assessment of arterial structure and function in patients with coarctation of the aorta undergoing stenting. Int J Cardiovasc Imaging. 2016 May;32(5):729-39. doi: 10.1007/s10554-015-0827-3. Epub 2016 Jan 2. PMID 26723574
- [Background] Thomas MN, Weninger E, Angele M, Bosch F, Pratschke S, Andrassy J, Rentsch M, Stangl M, Hartwig W, Werner J, Guba M. Intraoperative simulation of remnant liver function during anatomic liver resection with indocyanine green clearance (LiMON) measurements. HPB (Oxford). 2015 Jun;17(6):471-6. doi: 10.1111/hpb.12380. Epub 2015 Jan 8. PMID 25581073
- [Background] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Background] Peres A, Martins JD, Parames F, Gil R, Matias C, Franco J, Freitas I, Trigo C, Fragata J, Pinto FF. Isolated aortic coarctation: experience in 100 consecutive patients. Rev Port Cardiol. 2010 Jan;29(1):23-35. English, Portuguese. PMID 20391897
- [Background] Quennelle S, Powell AJ, Geva T, Prakash A. Persistent Aortic Arch Hypoplasia After Coarctation Treatment Is Associated With Late Systemic Hypertension. J Am Heart Assoc. 2015 Jun 25;4(7):e001978. doi: 10.1161/JAHA.115.001978. PMID 26112642
- [Background] Pedersen TA, Pedersen EB, Munk K, Hjortdal VE, Emmertsen K, Andersen NH. High pulse pressure is not associated with abnormal activation of the renin-angiotensin-aldosterone system in repaired aortic coarctation. J Hum Hypertens. 2015 Apr;29(4):268-73. doi: 10.1038/jhh.2014.75. Epub 2014 Aug 28. PMID 25355011
- [Background] Chen SS, Donald AE, Storry C, Halcox JP, Bonhoeffer P, Deanfield JE. Impact of aortic stenting on peripheral vascular function and daytime systolic blood pressure in adult coarctation. Heart. 2008 Jul;94(7):919-24. doi: 10.1136/hrt.2006.109389. Epub 2007 Aug 8. PMID 17686804
- [Background] Toro-Salazar OH, Steinberger J, Thomas W, Rocchini AP, Carpenter B, Moller JH. Long-term follow-up of patients after coarctation of the aorta repair. Am J Cardiol. 2002 Mar 1;89(5):541-7. doi: 10.1016/s0002-9149(01)02293-7. PMID 11867038
- [Background] Koller M, Rothlin M, Senning A. Coarctation of the aorta: review of 362 operated patients. Long-term follow-up and assessment of prognostic variables. Eur Heart J. 1987 Jul;8(7):670-9. doi: 10.1093/eurheartj/8.7.670. PMID 3653118
- [Background] Choudhary P, Canniffe C, Jackson DJ, Tanous D, Walsh K, Celermajer DS. Late outcomes in adults with coarctation of the aorta. Heart. 2015 Aug;101(15):1190-5. doi: 10.1136/heartjnl-2014-307035. Epub 2015 Mar 25. PMID 25810155
- [Background] Hoimyr H, Christensen TD, Emmertsen K, Johnsen SP, Riis A, Hansen OK, Hjortdal VE. Surgical repair of coarctation of the aorta: up to 40 years of follow-up. Eur J Cardiothorac Surg. 2006 Dec;30(6):910-6. doi: 10.1016/j.ejcts.2006.09.016. Epub 2006 Oct 23. PMID 17056267
- [Background] Mandalenakis Z, Rosengren A, Lappas G, Eriksson P, Hansson PO, Dellborg M. Ischemic Stroke in Children and Young Adults With Congenital Heart Disease. J Am Heart Assoc. 2016 Feb 23;5(2):e003071. doi: 10.1161/JAHA.115.003071. PMID 26908411
- [Background] Vogt M, Kuhn A, Baumgartner D, Baumgartner C, Busch R, Kostolny M, Hess J. Impaired elastic properties of the ascending aorta in newborns before and early after successful coarctation repair: proof of a systemic vascular disease of the prestenotic arteries? Circulation. 2005 Jun 21;111(24):3269-73. doi: 10.1161/CIRCULATIONAHA.104.529792. Epub 2005 Jun 13. PMID 15956120
- [Background] Li VW, Cheung YF. Arterial-left ventricular-left atrial coupling late after repair of aortic coarctation and interruption. Eur Heart J Cardiovasc Imaging. 2015 Jul;16(7):771-80. doi: 10.1093/ehjci/jeu309. Epub 2015 Jan 14. PMID 25588795
- [Background] Agnoletti G, Bonnet C, Bonnet D, Sidi D, Aggoun Y. Mid-term effects of implanting stents for relief of aortic recoarctation on systemic hypertension, carotid mechanical properties, intimal medial thickness and reflection of the pulse wave. Cardiol Young. 2005 Jun;15(3):245-50. doi: 10.1017/S1047951105000521. PMID 15865825
- [Background] Ou P, Celermajer DS, Jolivet O, Buyens F, Herment A, Sidi D, Bonnet D, Mousseaux E. Increased central aortic stiffness and left ventricular mass in normotensive young subjects after successful coarctation repair. Am Heart J. 2008 Jan;155(1):187-93. doi: 10.1016/j.ahj.2007.09.008. Epub 2007 Nov 19. PMID 18082512
- [Background] de Divitiis M, Pilla C, Kattenhorn M, Zadinello M, Donald A, Leeson P, Wallace S, Redington A, Deanfield JE. Vascular dysfunction after repair of coarctation of the aorta: impact of early surgery. Circulation. 2001 Sep 18;104(12 Suppl 1):I165-70. doi: 10.1161/hc37t1.094900. PMID 11568050
- [Background] Trojnarska O, Szczepaniak-Chichel L, Mizia-Stec K, Gabriel M, Bartczak A, Grajek S, Gasior Z, Kramer L, Tykarski A. Vascular remodeling in adults after coarctation repair: impact of descending aorta stenosis and age at surgery. Clin Res Cardiol. 2011 May;100(5):447-55. doi: 10.1007/s00392-010-0263-2. Epub 2010 Dec 16. PMID 21161708
- [Background] Brili S, Antonopoulos AS, Oikonomou E, Kalampogias A, Papamikroulis GA, Chrysochoou C, Mourouzis K, Nihoyanopoulos P, Tousoulis D. Impairment of arterial elastic properties and elevated circulating levels of transforming growth factor-beta in subjects with repaired coarctation of aorta. Int J Cardiol. 2016 Mar 15;207:282-3. doi: 10.1016/j.ijcard.2016.01.168. Epub 2016 Jan 11. No abstract available. PMID 26812641
- [Background] Moutafi AC, Alissafi T, Chamakou A, Chryssanthopoulos S, Thanopoulos V, Dellos C, Xanthou G, Tousoulis D, Stefanadis C, Gatzoulis MA, Davos CH. Neurohormonal activity and vascular properties late after aortic coarctation repair. Int J Cardiol. 2012 Sep 6;159(3):211-6. doi: 10.1016/j.ijcard.2011.02.071. Epub 2011 Mar 22. PMID 21429604
- [Background] Swan L, Kraidly M, Vonder Muhll I, Collins P, Gatzoulis MA. Surveillance of cardiovascular risk in the normotensive patient with repaired aortic coarctation. Int J Cardiol. 2010 Mar 18;139(3):283-8. doi: 10.1016/j.ijcard.2008.10.043. Epub 2008 Dec 6. PMID 19059656
- [Background] Barton CH, Ni Z, Vaziri ND. Enhanced nitric oxide inactivation in aortic coarctation-induced hypertension. Kidney Int. 2001 Sep;60(3):1083-7. doi: 10.1046/j.1523-1755.2001.0600031083.x. PMID 11532103
- [Background] Xu C, Lee S, Singh TM, Sho E, Li X, Sho M, Masuda H, Zarins CK. Molecular mechanisms of aortic wall remodeling in response to hypertension. J Vasc Surg. 2001 Mar;33(3):570-8. doi: 10.1067/mva.2001.112231. PMID 11241129
- [Background] Sarkola T, Redington AN, Slorach C, Hui W, Bradley T, Jaeggi E. Assessment of vascular phenotype using a novel very-high-resolution ultrasound technique in adolescents after aortic coarctation repair and/or stent implantation: relationship to central haemodynamics and left ventricular mass. Heart. 2011 Nov;97(21):1788-93. doi: 10.1136/hrt.2011.226241. Epub 2011 Jul 27. PMID 21795301
- [Background] Kutty S, Rangamani S, Venkataraman J, Li L, Schuster A, Fletcher SE, Danford DA, Beerbaum P. Reduced global longitudinal and radial strain with normal left ventricular ejection fraction late after effective repair of aortic coarctation: a CMR feature tracking study. Int J Cardiovasc Imaging. 2013 Jan;29(1):141-50. doi: 10.1007/s10554-012-0061-1. Epub 2012 May 12. PMID 22581073
- [Background] Lombardi KC, Northrup V, McNamara RL, Sugeng L, Weismann CG. Aortic stiffness and left ventricular diastolic function in children following early repair of aortic coarctation. Am J Cardiol. 2013 Dec 1;112(11):1828-33. doi: 10.1016/j.amjcard.2013.07.052. Epub 2013 Sep 13. PMID 24035164
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] LaDisa JF Jr, Bozdag S, Olson J, Ramchandran R, Kersten JR, Eddinger TJ. Gene Expression in Experimental Aortic Coarctation and Repair: Candidate Genes for Therapeutic Intervention? PLoS One. 2015 Jul 24;10(7):e0133356. doi: 10.1371/journal.pone.0133356. eCollection 2015. PMID 26207811
- [Background] Hager A, Bildau J, Kreuder J, Kaemmerer H, Hess J. Impact of genomic polymorphism on arterial hypertension after aortic coarctation repair. Int J Cardiol. 2011 Aug 18;151(1):63-8. doi: 10.1016/j.ijcard.2010.04.090. Epub 2010 Jun 7. PMID 20537417
- [Background] Niwa K, Perloff JK, Bhuta SM, Laks H, Drinkwater DC, Child JS, Miner PD. Structural abnormalities of great arterial walls in congenital heart disease: light and electron microscopic analyses. Circulation. 2001 Jan 23;103(3):393-400. doi: 10.1161/01.cir.103.3.393. PMID 11157691
- [Background] Yokoyama U, Ichikawa Y, Minamisawa S, Ishikawa Y. Pathology and molecular mechanisms of coarctation of the aorta and its association with the ductus arteriosus. J Physiol Sci. 2017 Mar;67(2):259-270. doi: 10.1007/s12576-016-0512-x. Epub 2016 Dec 20. PMID 28000176
- [Background] Ou P, Bonnet D, Auriacombe L, Pedroni E, Balleux F, Sidi D, Mousseaux E. Late systemic hypertension and aortic arch geometry after successful repair of coarctation of the aorta. Eur Heart J. 2004 Oct;25(20):1853-9. doi: 10.1016/j.ehj.2004.07.021. PMID 15474701
- [Background] Redheuil A, Yu WC, Wu CO, Mousseaux E, de Cesare A, Yan R, Kachenoura N, Bluemke D, Lima JA. Reduced ascending aortic strain and distensibility: earliest manifestations of vascular aging in humans. Hypertension. 2010 Feb;55(2):319-26. doi: 10.1161/HYPERTENSIONAHA.109.141275. Epub 2010 Jan 11. PMID 20065154
- [Background] Parker FB Jr, Streeten DH, Farrell B, Blackman MS, Sondheimer HM, Anderson GH Jr. Preoperative and postoperative renin levels in coarctation of the aorta. Circulation. 1982 Sep;66(3):513-4. doi: 10.1161/01.cir.66.3.513. PMID 7046989
- [Background] Roegel JC, Heinrich E, De Jong W, Stephan D, Charpentier A, Eisenmann B, Imbs JL. Vascular and neuroendocrine components in altered blood pressure regulation after surgical repair of coarctation of the aorta. J Hum Hypertens. 1998 Aug;12(8):517-25. doi: 10.1038/sj.jhh.1000666. PMID 9759985
- [Background] Beekman RH, Katz BP, Moorehead-Steffens C, Rocchini AP. Altered baroreceptor function in children with systolic hypertension after coarctation repair. Am J Cardiol. 1983 Jul;52(1):112-7. doi: 10.1016/0002-9149(83)90080-2. PMID 6858899
- [Background] Polson JW, McCallion N, Waki H, Thorne G, Tooley MA, Paton JF, Wolf AR. Evidence for cardiovascular autonomic dysfunction in neonates with coarctation of the aorta. Circulation. 2006 Jun 20;113(24):2844-50. doi: 10.1161/CIRCULATIONAHA.105.602748. Epub 2006 Jun 12. PMID 16769911
- [Background] Clarkson PM, Nicholson MR, Barratt-Boyes BG, Neutze JM, Whitlock RM. Results after repair of coarctation of the aorta beyond infancy: a 10 to 28 year follow-up with particular reference to late systemic hypertension. Am J Cardiol. 1983 May 15;51(9):1481-8. doi: 10.1016/0002-9149(83)90661-6. PMID 6846181
- [Background] Bhatt AB, Defaria Yeh D. Long-term outcomes in coarctation of the aorta: an evolving story of success and new challenges. Heart. 2015 Aug;101(15):1173-5. doi: 10.1136/heartjnl-2015-307641. Epub 2015 May 29. No abstract available. PMID 26025083
- [Background] Giordano U, Giannico S, Turchetta A, Hammad F, Calzolari F, Calzolari A. The influence of different surgical procedures on hypertension after repair of coarctation. Cardiol Young. 2005 Oct;15(5):477-80. doi: 10.1017/S1047951105001332. PMID 16164785
- [Background] Kenny D, Polson JW, Martin RP, Wilson DG, Caputo M, Cockcroft JR, Paton JF, Wolf AR. Surgical approach for aortic coarctation influences arterial compliance and blood pressure control. Ann Thorac Surg. 2010 Aug;90(2):600-4. doi: 10.1016/j.athoracsur.2010.04.098. PMID 20667357
- [Background] Bassareo PP, Marras AR, Manai ME, Mercuro G. The influence of different surgical approaches on arterial rigidity in children after aortic coarctation repair. Pediatr Cardiol. 2009 May;30(4):414-8. doi: 10.1007/s00246-008-9381-2. Epub 2009 Jan 30. PMID 19184170
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Townsend RR, Wilkinson IB, Schiffrin EL, Avolio AP, Chirinos JA, Cockcroft JR, Heffernan KS, Lakatta EG, McEniery CM, Mitchell GF, Najjar SS, Nichols WW, Urbina EM, Weber T; American Heart Association Council on Hypertension. Recommendations for Improving and Standardizing Vascular Research on Arterial Stiffness: A Scientific Statement From the American Heart Association. Hypertension. 2015 Sep;66(3):698-722. doi: 10.1161/HYP.0000000000000033. Epub 2015 Jul 9. No abstract available. PMID 26160955
- [Background] Ibrahim el-SH, Johnson KR, Miller AB, Shaffer JM, White RD. Measuring aortic pulse wave velocity using high-field cardiovascular magnetic resonance: comparison of techniques. J Cardiovasc Magn Reson. 2010 May 11;12(1):26. doi: 10.1186/1532-429X-12-26. PMID 20459799
- [Background] Grotenhuis HB, Westenberg JJ, Steendijk P, van der Geest RJ, Ottenkamp J, Bax JJ, Jukema JW, de Roos A. Validation and reproducibility of aortic pulse wave velocity as assessed with velocity-encoded MRI. J Magn Reson Imaging. 2009 Sep;30(3):521-6. doi: 10.1002/jmri.21886. PMID 19711407
- [Background] Huybrechts SA, Devos DG, Vermeersch SJ, Mahieu D, Achten E, de Backer TL, Segers P, van Bortel LM. Carotid to femoral pulse wave velocity: a comparison of real travelled aortic path lengths determined by MRI and superficial measurements. J Hypertens. 2011 Aug;29(8):1577-82. doi: 10.1097/HJH.0b013e3283487841. PMID 21666491
- [Background] Lerman A, Zeiher AM. Endothelial function: cardiac events. Circulation. 2005 Jan 25;111(3):363-8. doi: 10.1161/01.CIR.0000153339.27064.14. No abstract available. PMID 15668353
- [Background] Selamet Tierney ES, Newburger JW, Gauvreau K, Geva J, Coogan E, Colan SD, de Ferranti SD. Endothelial pulse amplitude testing: feasibility and reproducibility in adolescents. J Pediatr. 2009 Jun;154(6):901-5. doi: 10.1016/j.jpeds.2008.12.028. Epub 2009 Feb 12. PMID 19217124
- [Background] Kelly R, Fitchett D. Noninvasive determination of aortic input impedance and external left ventricular power output: a validation and repeatability study of a new technique. J Am Coll Cardiol. 1992 Oct;20(4):952-63. doi: 10.1016/0735-1097(92)90198-v. PMID 1527307
- [Background] Singh JP, Larson MG, Manolio TA, O'Donnell CJ, Lauer M, Evans JC, Levy D. Blood pressure response during treadmill testing as a risk factor for new-onset hypertension. The Framingham heart study. Circulation. 1999 Apr 13;99(14):1831-6. doi: 10.1161/01.cir.99.14.1831. PMID 10199879
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Background] Cooke JP. Asymmetrical dimethylarginine: the Uber marker? Circulation. 2004 Apr 20;109(15):1813-8. doi: 10.1161/01.CIR.0000126823.07732.D5. No abstract available. PMID 15096461
- [Background] Kannel WB, Gordon T, Offutt D. Left ventricular hypertrophy by electrocardiogram. Prevalence, incidence, and mortality in the Framingham study. Ann Intern Med. 1969 Jul;71(1):89-105. doi: 10.7326/0003-4819-71-1-89. No abstract available. PMID 4239887
- [Background] Lloyd-Jones DM, Hong Y, Labarthe D, Mozaffarian D, Appel LJ, Van Horn L, Greenlund K, Daniels S, Nichol G, Tomaselli GF, Arnett DK, Fonarow GC, Ho PM, Lauer MS, Masoudi FA, Robertson RM, Roger V, Schwamm LH, Sorlie P, Yancy CW, Rosamond WD; American Heart Association Strategic Planning Task Force and Statistics Committee. Defining and setting national goals for cardiovascular health promotion and disease reduction: the American Heart Association's strategic Impact Goal through 2020 and beyond. Circulation. 2010 Feb 2;121(4):586-613. doi: 10.1161/CIRCULATIONAHA.109.192703. Epub 2010 Jan 20. PMID 20089546
- [Background] Verma S, Siu SC. Aortic dilatation in patients with bicuspid aortic valve. N Engl J Med. 2014 May 15;370(20):1920-9. doi: 10.1056/NEJMra1207059. No abstract available. PMID 24827036
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Background] Quaal SJ. Interpreting the arterial pressure waveform in the intra-aortic balloon-pumped patient. Prog Cardiovasc Nurs. 2001 Summer;16(3):116-8, 125. doi: 10.1111/j.0889-7204.2001.00591.x. PMID 11464433
- [Background] Walhout RJ. Assessment of proximal and distal aortic properties with magnetic resonance after successful coarctation management in adults. Advances in the management and surveillance of patients with aortic coarctation. 2009/06/26 ed: Universiteit Amsterdam; 2009. p. 122-30.
- [Background] Colan SD. Normal echocardiographic values for cardiovascular structures. In: Lai WW, Cohen MS, Geva T, Mertens L, editors. Echocardiography in Pediatric and Congenital Heart Disease. West Sussex, UK: Wiley-Blackwell; 2009. p. Appendix 1, pp 765-85.
- [Derived] Martins JD, Zachariah J, Selamet Tierney ES, Truong U, Morris SA, Kutty S, de Ferranti SD, Guarino M, Thomas B, Oliveira D, Marinho A, Antonio M, Gauvreau K, Jalles N, Geva T, Carmo MM, Prakash A; LOVE-COARCT Study. Impact of Treatment Modality on Vascular Function in Coarctation of the Aorta: The LOVE - COARCT Study. J Am Heart Assoc. 2019 Apr 2;8(7):e011536. doi: 10.1161/JAHA.118.011536. PMID 30929556